CLINICAL TRIAL: NCT03451266
Title: Effects of Vitamin C Administration on Extravascular Lung Water in Patients With Severe Features of Preeclampsia: a Randomized, Placebo-controlled Trial
Brief Title: Effects of Vitamin C Administration on Extravascular Lung Water in Patients With Severe Features of Preeclampsia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, Principal Investigator, Head of the Perinatal Intensive Medicine Unit, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017 0031
Record Dates: First submitted 2018-02-17; First posted 2018-03-01 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Preeclampsia Severe; Preeclampsia Postpartum
Keywords: preeclampsia; vitamin C; lung ultrasound
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): 1,5g of IV vitamin C in 100 ml 0.9% NaCl within 30 min of delivery and then every 6 hours for the first 72 hours post-partum (vitamin C arm).
  Interventions: Drug: Vitamin C
- placebo (Placebo Comparator): 100 ml of IV 0.9% NaCl within 30 min of delivery and then every 6 hours for the first 72 hours post-partum (placebo arm).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin C — 1,5g of IV vitamin C in 100 ml 0.9% NaCl within 30 min of delivery and then every 6 hours for the first 72 hours post-partum.
  Arms: Vitamin C
Drug: placebo — 100 ml of IV 0.9% NaCl within 30 min of delivery and then every 6 hours for the first 72 hours post-partum.
  Arms: placebo

SUMMARY:
The objective of the study is to determine whether administration of vitamin C (1.5g/6 hours) in the first three days post-partum reduces the amount of extravascular lung water assessed by lung ultrasound in patients with severe preeclampsia.

DETAILED DESCRIPTION:
Risk of fluid over-resuscitation is high in preeclampsia due to endothelial dysfunction and resulting increased vascular permeability. The Confidential Enquiry into Maternal Deaths in the UK reported six maternal deaths between 1994 and 1996 due to adult respiratory distress syndrome (ARDS) that appeared to be related to poor fluid management in women with preeclampsia. On the basis of these reported deaths, recommendations on limiting intravenous fluids to not more than to 80 ml/hour (or 1 ml/kg/h) have been made. Nevertheless, preeclampsia remains the leading cause of pulmonary edema in the peripartum period. Moreover, in some preeclamptic patients higher rates of intravenous fluid administration may be necessary to adequately correct tissue hypoperfusion.

Zieleskiewicz et al. were the first to demonstrate that lung ultrasound (LUS) can be used to objectively evaluate increased extravascular lung water (EVLW) in patients with preeclampsia. Ambrozic et al. recently confirmed these results and showed that the amount of EVLW assessed by LUS is increased in preeclamptic patients compared to healthy controls and that it decreases rapidly in the first four days following delivery.

It has been reported that administration of high-dose ascorbic acid (vitamin C) reduces vascular permeability in animals. In 2000, Tanaka et al. reported an RCT involving 37 patients with major burns (>30% body surface area) randomized regarding whether or not to receive an infusion of IV vitamin C, 66 mg/kg/h for the first 24 hours of hospitalization. Patients in the vitamin C group required less fluid resuscitation, had higher urine output, and developed less wound edema. This translated into improved oxygenation and less time on mechanical ventilation among the vitamin C group (average of 12 vs. 21 days of ventilation, p=0.03). In 2002, Nathens et al. randomized patients shortly after admission to a surgical ICU to no therapy vs. a combination of enteral vitamin E plus IV vitamin C 1000 mg/8h until ICU discharge. The primary endpoint was a composite of pneumonia or ARDS. Although there were trends towards fewer pulmonary complications among patients treated with antioxidants, these did not reach statistical significance (the study was underpowered due to low rates of respiratory complications). However, patients treated with vitamins E and C fared better on a variety of secondary endpoints including less time on the ventilator and less multiorgan failure.

In women with established preeclampsia, there is evidence of oxidative stress and decreased concentrations of vitamin C. An initial RCT on prophylactic supplementation with oral antioxidants, including 1g vitamin C daily, showed a significant reduction in preeclampsia (8 percent vs. 17 percent) in high-risk pregnancies. Subsequent large RCTs have, however, reported no significant reduction in the risks of preeclampsia, intrauterine growth restriction, or the risk of death or other serious outcomes in infants associated with oral vitamin C supplementation.There are no studies to date on use of higher dose IV vitamin C administration for reduction of capillary leak and consequently EVLW in patients with severe forms of preeclampsia. Given the safety (see below) and low costs of vitamin C this could be a promising approach to increase fluid tolerance in these patients. If vitamin C reduces vascular permeability in preeclampsia patients to the same degree that it seems to reduce vascular permeability in other conditions, such as burns, it could reduce the risk of pulmonary complications associated with this disease. At the same time, vitamin C therapy could allow safe additional fluid administration in patients with preeclampsia who are fluid responsive and in whom further increases in preload would be beneficial for preventing end-organ damage such as pre-renal acute kidney injury.

Safety of vitamin C

Safety of vitamin C has been well established even at high doses. For example, none of the above studies reported any adverse event, despite the use of very high doses by Tanaka et al. (1.6 grams/kg over 24 hours). One potential concern regarding vitamin C is that it may be metabolized into oxalic acid, leading to calcium oxalate nephropathy. This doesn't seem to be a significant problem for several reasons:

* Oxalate formation is a dose-dependent toxicity. This has rarely been reported from short courses of IV vitamin C, but only at much higher doses (>40 grams/day).
* In 2014, Fowler et al. published a phase I safety trial of vitamin C in patients with severe sepsis. Their prospective RCT involved patients with severe sepsis in a medical ICU. 24 patients were randomized to receive placebo, low-dose vitamin C (12.5 mg/kg IV/6hr), or high-dose vitamin C (50 mg/kg IV/6hr). The primary endpoint was safety and tolerability, with no adverse events noted.
* Recently Marik et al. published a before-after study investigating the impact of treating sepsis with a combination of thiamine 200 mg IV/12hr, Vitamin C 1.5 g/6hr, and hydrocortisone 50 mg IV/6hr. Mortality was substantially reduced in patients receiving vitamin C (p<0.001). Moreover, vitamin C use correlated with improved renal outcomes (the rate of dialysis was reduced from 33% to 10%, p=0.02).

Another concern which has been raised is that vitamin C at extremely high doses may have a pro-oxidant effect. This was shown not to occur even at a dose of 7.5 grams IV daily.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnancy with severe featutes of preeclampsia (any of the following):

* Systolic blood pressure of 160 mm Hg or higher, or diastolic blood pressure of 110 mm Hg or higher on two occasions at least 4 hours apart while the patient is on bed rest (unless antihypertensive therapy is initiated before this time)
* Thrombocytopenia (platelet count less than 100x109/L)
* Impaired liver function as indicated by abnormally elevated blood concentrations of liver enzymes (to twice normal concentration), severe persistent right upper quadrant or epigastric pain unresponsive to medication and not accounted for by alternative diagnoses, or both
* Progressive renal insufficiency (serum creatinine concentration greater 97 µmol/L or a doubling of the serum creatinine concentration in the absence of other renal disease)
* Pulmonary edema
* New-onset cerebral or visual disturbances

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Echo Comet Score at day 1 post-delivery | Echo Comet Score (ECS) will be assessed by lung ultrasound at day 1 following delivery
  The primary outcome studied will be the Echo Comet Score (ECS) at day 1 following delivery in the vitamin C vs. placebo group. ECS will be obtained by the 28-rib interspaces technique dividing the chest wall in 12 areas on the left (from the second to the fourth intercostal space) and 16 areas on the right (from the second to the fifth intercostal space) anterior and lateral hemithorax. The sum of ultrasonographic B-lines found on each scanning site (from 0 to 10) will yield a score ranging from 0 to 280. ECS denotes the amount of extravascular fluid in the lung, i.e. the higher the ESC, the larger the amount of extravascular lung water.

SECONDARY OUTCOMES:
Echo Comet Score at day 2 post-delivery | Echo Comet Score (ECS) will be assessed by lung ultrasound at day 2 following delivery
  One of the secondary outcomes studied will be the Echo Comet Score (ECS) at day 2 following delivery in the vitamin C vs. placebo group. ECS will be obtained by the 28-rib interspaces technique dividing the chest wall in 12 areas on the left (from the second to the fourth intercostal space) and 16 areas on the right (from the second to the fifth intercostal space) anterior and lateral hemithorax. The sum of ultrasonographic B-lines found on each scanning site (from 0 to 10) will yield a score ranging from 0 to 280. ECS denotes the amount of extravascular fluid in the lung, i.e. the higher the ESC, the larger the amount of extravascular lung water.
Echo Comet Score at day 3 post-delivery | Echo Comet Score (ECS) will be assessed by lung ultrasound at day 3 following delivery
  One of the secondary outcomes studied will be the Echo Comet Score (ECS) at day 3 following delivery in the vitamin C vs. placebo group. ECS will be obtained by the 28-rib interspaces technique dividing the chest wall in 12 areas on the left (from the second to the fourth intercostal space) and 16 areas on the right (from the second to the fifth intercostal space) anterior and lateral hemithorax. The sum of ultrasonographic B-lines found on each scanning site (from 0 to 10) will yield a score ranging from 0 to 280. ECS denotes the amount of extravascular fluid in the lung, i.e. the higher the ESC, the larger the amount of extravascular lung water.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zieleskiewicz L, Contargyris C, Brun C, Touret M, Vellin A, Antonini F, Muller L, Bretelle F, Martin C, Leone M. Lung ultrasound predicts interstitial syndrome and hemodynamic profile in parturients with severe preeclampsia. Anesthesiology. 2014 Apr;120(4):906-14. doi: 10.1097/ALN.0000000000000102. PMID 24694847
- [Background] Ambrozic J, Brzan Simenc G, Prokselj K, Tul N, Cvijic M, Lucovnik M. Lung and cardiac ultrasound for hemodynamic monitoring of patients with severe pre-eclampsia. Ultrasound Obstet Gynecol. 2017 Jan;49(1):104-109. doi: 10.1002/uog.17331. Epub 2016 Dec 1. PMID 27736042
- [Background] Matsuda T, Tanaka H, Hanumadass M, Gayle R, Yuasa H, Abcarian H, Matsuda H, Reyes H. Effects of high-dose vitamin C administration on postburn microvascular fluid and protein flux. J Burn Care Rehabil. 1992 Sep-Oct;13(5):560-6. doi: 10.1097/00004630-199209000-00009. PMID 1452590
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Derived] Korenc M, Zieleskiewicz L, Stopar Pintaric T, Blajic I, Ambrozic J, Lucovnik M. The effect of vitamin C on pulmonary oedema in patients with severe preeclampsia: A single-centre, randomised, placebo-controlled, double-blind trial. Anaesth Crit Care Pain Med. 2021 Feb;40(1):100800. doi: 10.1016/j.accpm.2021.100800. Epub 2021 Jan 14. PMID 33453456

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03451266/Prot_SAP_000.pdf